CLINICAL TRIAL: NCT05341895
Title: The Effect of Kinesiotape Applied on Paraspinal Muscles on Balance in Individuals With Multiple Sclerosis
Brief Title: Kinesiotape on Balance in With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Furkan BİLEK, Lecturer, Firat University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Firat Un.
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Individuals With Multiple Sclerosis; With Ataxia Symptoms; No Secondary Disease Affecting Balance
Keywords: Multiple Sclerosis; Balance; Ataxia; Kinesiotape
MeSH Terms: conditions — Multiple Sclerosis; Ataxia | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: prospective
Masking Description: The patient does not know the purpose of the kinesiotape
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotape (Other): Kinesiotape applied to the paraspinal muscles
  Interventions: Other: Kinesiotape
- Placebo (No Intervention): No intervention

INTERVENTIONS:
Other: Kinesiotape — Taping
  Arms: kinesiotape

SUMMARY:
Multiple Sclerosis (MS), a chronic inflammatory disease of the central nervous system, is a disease characterized by myelin, oligodendrocyte and axon damage. Research continues on the autoimmune, infectious, environmental, vascular and genetic origins of this disease, which affects approximately 2.5 million people in the world and is seen 2-3 times more in women than in men. Although the signs and symptoms of the disease vary according to the location of the lesion; frequently, loss of strength, spasticity, sensory disturbances, fatigue, ataxia, autonomic dysfunction, and decreased visual acuity are observed. With these approaches, the effect of Kinesiotape application on balance will be investigated in individuals with ataxic MS. Based on this idea, our work; It was planned to investigate the effect of kinesiotape application on balance in individuals diagnosed with ataxic multiple sclerosis.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS), a chronic inflammatory disease of the central nervous system, is a disease characterized by myelin, oligodendrocyte and axon damage. Research continues on the autoimmune, infectious, environmental, vascular and genetic origins of this disease, which affects approximately 2.5 million people in the world and is seen 2-3 times more in women than in men. Although the signs and symptoms of the disease vary according to the location of the lesion; frequently, loss of strength, spasticity, sensory disturbances, fatigue, ataxia, autonomic dysfunction, and decreased visual acuity are observed.

Balance problems are seen in 50-80% of MS patients. Balance requires the controlled coordination of many central nervous system structures. Integration of vestibular, visual and somatosensory information is required to achieve and maintain balance. Vestibular ataxia occurs as a result of problems in the vestibular systems. These patients try to reduce head and eye movements as much as possible in order to maintain their balance. Symptoms arising from vestibular system dysfunction are seen in 49-59% of MS patients. symptoms; includes vertigo, drowsiness, and balance disorder. Somatosensory problems are seen in 80% of MS patients. Since the somatosensory system is one of the most fundamental factors in maintaining postural control and balance, sensory ataxia findings are frequently encountered in these patients due to the somatosensory system involvement. The most basic finding seen in these patients is that they perform many activities in daily life mostly using the visual system, since the information coming from the somatosensory system is not sufficient. The cerebellum and its efferent and afferent pathways are commonly affected in MS; and cerebellar ataxia is one of the most common symptoms especially in the progressive phase of the disease. Gait ataxia is thought to occur predominantly due to damage to the anterior lobe of the cerebellum. Trunk, extremity, or gait ataxia findings may occur singly and/or together, depending on the affected area of the cerebellum. balance dysfunction in MS patients; It is shaped mainly on the basis of three problems: decreased ability to maintain the existing position, a slow and limited movement towards the limits of stability, and delayed responses to postural displacements. In MS patients, functional balance performance is also affected in situations that require multitasking.

Kinesiotape is a relatively new method used in rehabilitation programs, and it is increasingly becoming an adjunctive treatment option for multidisciplinary rehabilitation in MS patients. It is a thin and elastic band that can stretch up to 120-140% of its original length. It is therefore highly elastic and causes fewer mechanism restrictions compared to the conventional tape. This technique normalizes muscle function, increases lymphatic and vascular flow, reduces pain, strengthens weakened muscles, and helps with postural alignment by relaxing overused muscles. It has been claimed that the effects of kinesiotape may result from sensorimotor and proprioceptive feedback mechanisms. Kinesiotape provides rapid sensorimotor feedback: patients usually report relief of symptoms, increased comfort level, or stability of the involved joint within a few days. Kinesiotape may be an alternative rehabilitation option when a rapid effect is required in the treatment of MS. However, more clinical and neurophysiological studies are needed to clarify the mechanism of action and effects of the Kinesiotape technique.

With these approaches, the effect of Kinesiotape application on balance will be investigated in individuals with ataxic MS. Based on this idea, our work; It was planned to investigate the effect of kinesiotape application on balance in individuals diagnosed with ataxic multiple sclerosis.

In our study, patients diagnosed with MS by a neurologist at Fırat University Hospital will be evaluated.

From patient records, demographic characteristics; patients' age, gender, body weight, height, EDSS score, occupation and educational status, history of the disease; The MS type will be registered. To our neurological evaluation form; reflexes, sensory defects, cranial nerve lesion, visual disturbances, speech problems, balance and functional status will be obtained.

With these data, the effects of Kinesiotape application on the balance status of patients will be investigated.

Functional Reach Test, Timed Get Up and Go Test, 25 Steps Walk Test, 3 Meter backward walking Test and Win-Track walking platform evaluation data will be taken from the participants.

Statistical analyzes of the study will be done with "Statistical Package for Social Sciences" (SPSS) Version IBM Statistic 20. Demographic data will be given as mean ± SD. Students t test will be used in continuous variables analysis and Chi-square test will be used in comparison of percentages. Differences below a P value <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* with ataxia symptoms with a diagnosis of multiple sclerosis No attacks in the last 3 months

Exclusion Criteria:

* Having other illnesses that may affect the balance allergic to kinesiotape

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-04-22 (Estimated); Study Completion 2022-05-06 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go Test | 1 week
  It is applied to evaluate the balance and fall risk of individuals. The patient is first asked to sit leaning on the chair. The patient is then asked to stand up, walk with regular steps for a predetermined distance of 3 meters, return at the end of 3 meters and sit in a chair. During the test, the patient's walking time is recorded in seconds with a stopwatch. The test was repeated three times and the mean value will be recorded
Win-Track Analysis | 1 week
  With the pressure measurement platform, static and dynamic pressure distributions, motion cycles, pressure, power, time and step parameters, as well as gait symmetry analysis data will be taken from the system
3-meter Backward walk Test | 1 week
  The 3-meter distance is marked with a black tape and participants are asked to align their heels with the black tape. Individuals are asked to walk backwards as soon as possible with the "walk" command and stop when they reach 3 meters. Meanwhile, the elapsed time is recorded in seconds. Evaluation will be done three times and the average time will be recorded

SECONDARY OUTCOMES:
Functional Reach Test | 1 week
  The FRT is a clinical assessment tool of balance and requires only a flattened measuring stick attached to the wall at the height of the participant's right acromion. In the test, a participant stands comfortably with their feet approximately shoulder-width apart and positions their preferred arm closest to the wall at 90° shoulder flexion. They reach as far as possible without falling and stepping. The examiner records the position of the distal ends of the finger in the starting position and the ending position, and the distance is the difference between the two positions, measured in cm
Timed 25-Foot Walk | 1 week
  The 25-Step Walking Test is a test that measures lower extremity functions. It has been developed for the purpose of recording the patient with this test at each examination. The patient is asked to walk in a predetermined interval. The average of both times is taken by noting the number of seconds spent on the way out and on the way back

CONTACTS AND LOCATIONS:
Overall Officials: Caner F Demir, MD professor, Principal Investigator — Firat University
Locations (2):
- Turkey (Türkiye) (2):
  - Furkan Bilek, Elâzığ
  - Fırat university, Elâzığ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frohman EM, Racke MK, Raine CS. Multiple sclerosis--the plaque and its pathogenesis. N Engl J Med. 2006 Mar 2;354(9):942-55. doi: 10.1056/NEJMra052130. No abstract available. PMID 16510748
- [Background] Mazumder R, Murchison C, Bourdette D, Cameron M. Falls in people with multiple sclerosis compared with falls in healthy controls. PLoS One. 2014 Sep 25;9(9):e107620. doi: 10.1371/journal.pone.0107620. eCollection 2014. PMID 25254633
- [Background] Marsden J, Pavlou M, Dennett R, Gibbon A, Knight-Lozano R, Jeu L, Flavell C, Freeman J, Bamiou DE, Harris C, Hawton A, Goodwin E, Jones B, Creanor S. Vestibular rehabilitation in multiple sclerosis: study protocol for a randomised controlled trial and cost-effectiveness analysis comparing customised with booklet based vestibular rehabilitation for vestibulopathy and a 12 month observational cohort study of the symptom reduction and recurrence rate following treatment for benign paroxysmal positional vertigo. BMC Neurol. 2020 Nov 27;20(1):430. doi: 10.1186/s12883-020-01983-y. PMID 33243182
- [Background] Jamali A, Sadeghi-Demneh E, Fereshtenajad N, Hillier S. Somatosensory impairment and its association with balance limitation in people with multiple sclerosis. Gait Posture. 2017 Sep;57:224-229. doi: 10.1016/j.gaitpost.2017.06.020. Epub 2017 Jun 24. PMID 28667904
- [Background] D'Ambrosio A, Pagani E, Riccitelli GC, Colombo B, Rodegher M, Falini A, Comi G, Filippi M, Rocca MA. Cerebellar contribution to motor and cognitive performance in multiple sclerosis: An MRI sub-regional volumetric analysis. Mult Scler. 2017 Aug;23(9):1194-1203. doi: 10.1177/1352458516674567. Epub 2016 Oct 19. PMID 27760859
- [Background] Cameron MH, Lord S. Postural control in multiple sclerosis: implications for fall prevention. Curr Neurol Neurosci Rep. 2010 Sep;10(5):407-12. doi: 10.1007/s11910-010-0128-0. PMID 20567946
- [Background] Yoshida A, Kahanov L. The effect of kinesio taping on lower trunk range of motions. Res Sports Med. 2007 Apr-Jun;15(2):103-12. doi: 10.1080/15438620701405206. PMID 17578750
- [Background] Kesselring J, Beer S. Symptomatic therapy and neurorehabilitation in multiple sclerosis. Lancet Neurol. 2005 Oct;4(10):643-52. doi: 10.1016/S1474-4422(05)70193-9. PMID 16168933
- [Background] Fu TC, Wong AM, Pei YC, Wu KP, Chou SW, Lin YC. Effect of Kinesio taping on muscle strength in athletes-a pilot study. J Sci Med Sport. 2008 Apr;11(2):198-201. doi: 10.1016/j.jsams.2007.02.011. Epub 2007 Jun 27. PMID 17588814
- [Background] Halseth T, McChesney JW, Debeliso M, Vaughn R, Lien J. The effects of kinesio taping on proprioception at the ankle. J Sports Sci Med. 2004 Mar 1;3(1):1-7. eCollection 2004 Mar. PMID 24497814
- [Background] Lin JJ, Hung CJ, Yang PL. The effects of scapular taping on electromyographic muscle activity and proprioception feedback in healthy shoulders. J Orthop Res. 2011 Jan;29(1):53-7. doi: 10.1002/jor.21146. PMID 20607815
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Goodman AD, Cohen JA, Cross A, Vollmer T, Rizzo M, Cohen R, Marinucci L, Blight AR. Fampridine-SR in multiple sclerosis: a randomized, double-blind, placebo-controlled, dose-ranging study. Mult Scler. 2007 Apr;13(3):357-68. doi: 10.1177/1352458506069538. Epub 2007 Jan 29. PMID 17439905
- [Background] Bilek F, Demir CF. Validity and reliability of the 3-meter backward walk test in mildly disabled persons with multiple sclerosis. Mult Scler Relat Disord. 2022 Feb;58:103532. doi: 10.1016/j.msard.2022.103532. Epub 2022 Jan 19. PMID 35066275
- [Background] Soke F, Eldemir S, Ozkan T, Ozkul C, Ozcan Gulsen E, Gulsen C, Eldemir K, Irkec C, Bilge Gonenli K, Batur Caglayan HZ, Guclu-Gunduz A. The functional reach test in people with multiple sclerosis: a reliability and validity study. Physiother Theory Pract. 2022 Nov;38(13):2905-2919. doi: 10.1080/09593985.2021.1938308. Epub 2021 Jun 17. PMID 34137673
- [Background] Ramachandra P, Maiya AG, Kumar P. Test-retest reliability of the Win-Track platform in analyzing the gait parameters and plantar pressures during barefoot walking in healthy adults. Foot Ankle Spec. 2012 Oct;5(5):306-12. doi: 10.1177/1938640012457680. Epub 2012 Sep 5. PMID 22956663